CLINICAL TRIAL: NCT01362231
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GS-6624 in Adult Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: A Study to Evaluate the Safety and Efficacy of GS-6624 (Formerly AB0024) in Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AB0024-201; NCT01242189 (obsolete NCT alias)
Record Dates: First submitted 2011-04-12; First posted 2011-05-30 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Fibrosis; Pulmonary Fibrosis; Lung Diseases; Interstitial
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Fibrosis; Pulmonary Fibrosis; Lung Diseases | interventions — simtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GS-6624 125mg (Experimental)
  Interventions: Drug: GS-6624
- Experimental: GS-6624 200mg (Experimental)
  Interventions: Drug: GS-6624

INTERVENTIONS:
Drug: GS-6624 — Patients will be treated with GS-6624 (125 or 200 mg) administered IV over 1 hour on specific days during the treatment period.
  Other Names: AB0024

SUMMARY:
The study consists of 2 parts: Part A is a randomized, multiple-dose, double-blind, placebo-controlled sequential dose escalation study to evaluate GS-6624 in subjects with Idiopathic Pulmonary Fibrosis (IPF) and was completed in October 2011.

Part B is a randomized, two-dose, open-label dose expansion study to evaluate GS-6624 in subjects with IPF and is currently enrolling.

DETAILED DESCRIPTION:
The primary objective of this study is to characterize the safety, tolerability, and PK of GS-6624 after multiple IV administrations in patients with IPF. The secondary objectives are to evaluate the formation of anti-GS-6624 antibodies and to measure the effects of GS-6624 on FVC, DLCO, and SGRQ score. A total of 48 patients will be enrolled. In the double-blind phase (Part A), a total of 18 patients were enrolled at 3 dose levels. Part A was completed in October 2011.

In Part B, 30 patients will be enrolled at 2 dose levels. Part B is open-label and is currently enrolling.

ELIGIBILITY:
Inclusion Criteria:

1. Acceptable results on pulmonary function tests
2. At rest oxygen saturation ≥90% on room air
3. Adequate organ function

Exclusion Criteria:

1. High resolution computer tomography pattern showing emphysema that is greater than fibrosis
2. Acceptable results on whole body plethysmography
3. History of clinically significant hepatic or renal disease
4. Poorly controlled or severe diabetes mellitus
5. Use of systemic immunosuppressants within 28 days of GS-6624 infusion

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To characterize the safety, tolerability, and pharmacokinetics (PK) of GS-6624 | 113 days
  To characterize the safety, tolerability, and pharmacokinetics (PK) of GS-6624 after multiple intravenous (IV) administrations in subjects with idiopathic pulmonary fibrosis (IPF).

SECONDARY OUTCOMES:
- To evaluate the formation of anti-GS-6624 antibodies. - To assess the effects of GS-6624 treatment on force vital capacity (FVC) and carbon dioxide diffusing capacity (DLCO) - To assess the effects of GS-6624 treatment on SGRQ | 113 Days
  Secondary Endpoints:
  * Anti-GS-6624 antibody formation;
  * Change in FVC and DLCO;
  * Change in SGRQ score.

CONTACTS AND LOCATIONS:
Overall Officials: Zung Thai, MD, Study Director — Gilead Sciences
Locations (7):
- United States (7):
  - Arizona Pulmonary Specialists, Scottsdale, Arizona
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Loess Hills Clinical Research Center, Council Bluffs, Iowa
  - UPMC Translational Research Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee